CLINICAL TRIAL: NCT01685138
Title: A Phase II, Multicenter, Single-arm Study of Oral LDK378 in Crizotinib naïve Adult Patients With ALK-activated Non-small Cell Lung Cancer
Brief Title: LDK378 in Crizotinib naïve Adult Patients With ALK-activated Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A2203; 2012-003474-36 (EudraCT Number)
Record Dates: First submitted 2012-09-04; First posted 2012-09-14 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Non small cell lung carcinoma; NSCLC; ALK; LDK378; Ceritinib; crizotinib naïve adult patients; ALK-activated non-small cell lung cancer; treatment of lung cancer after first metastasis; lung cancer; lung adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LDK378 (Ceritinib) (Experimental): Participants on this arm took oral LDK378 750 mg once daily.
  Interventions: Drug: LDK378

INTERVENTIONS:
Drug: LDK378 — LDK378/Ceritinib was supplied as 150 mg hard gelatin capsules and administered orally
  Other Names: Ceritinib

SUMMARY:
A single-arm, open-label, two-stage multicenter, phase II study. Patients were pre-screened for ALK positive status. Treatment with LDK378 at 750 mg qd was continued until the patient experienced unacceptable toxicity that precluded further treatment, discontinued treatment at the discretion of the investigator or patient, started a new anticancer therapy and/or died. LDK378 was continued beyond RECIST defined progressive disease (PD) as assessed by the investigator, if in the judgment of the investigator, there was evidence of clinical benefit. Patients who discontinued the study medication in the absence of progression continued to be followed for tumor assessment until the time of PD as assessed by the investigator. Male and female patients aged 18 or over with ALK-rearranged non-small cell cancer (NSCLC) were screened for eligibility. Patients had to have received no prior crizotinib, and had to be chemotherapy-naïve or been pretreated with cytotoxic chemotherapy (up to three prior lines).

ELIGIBILITY:
Key Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of stage IIIB or IV NSCLC that carried an ALK rearrangement, as per the FDA-approved Vysis ALK break-apart FISH assay (Abbott Molecular Inc.)
* Age 18 years or older at the time of informed consent.
* Patients must have NSCLC that had progressed during or after the last chemotherapy regimen received prior to the first dose of LDK378, if chemotherapy was received
* Patients must have been chemotherapy-naive or had received 1-3 lines of cytotoxic chemotherapy to treat their locally advanced or metastatic NSCLC
* Patients must have had a tumor tissue sample available, collected either at the time of diagnosis of NSCLC or any time since.
* Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 2, except for patients with grade 2 nausea/vomiting and/or grade 2 diarrhea despite optimal supportive therapy who were not allowed to participate in the study.

Key Exclusion criteria:

* Prior treatment with crizotinib, or any other ALK inhibitor investigational agent, for NSCLC
* Patients with known hypersensitivity to any of the excipients of LDK378.
* Patients with symptomatic central nervous system (CNS) metastases who were neurologically unstable or had required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms.
* History of carcinomatous meningitis.
* Presence or history of a malignant disease other than NSCLC that has been diagnosed and/or required therapy within the past 3 years.
* Clinically significant, uncontrolled heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (47):
- United States (4):
  - Massachusetts General Hospital Mass Gen 5, Boston, Massachusetts
  - Washington University School of Medicine Washington University (16), St Louis, Missouri
  - Sarah Cannon Research Institute Drug Ship - 4, Nashville, Tennessee
  - U of TX Southwestern Medical Center - SimmonsCompCancerCtr Clinical Research Office, Dallas, Texas
- Australia (2):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Franston, Victoria
- Belgium (2):
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Leuven
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Novartis Investigative Site, Saint-Herblain, France
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (5):
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Orbassano, TO
- Japan (8):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Sunto Gun, Shizuoka
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo
- Novartis Investigative Site, Auckland, New Zealand
- Novartis Investigative Site, Oslo, Norway
- Russia (3):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- South Korea (3):
  - Novartis Investigative Site, Seoul, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Stockholm, Sweden
- Taiwan (4):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
- United Kingdom (2):
  - Novartis Investigative Site, Colchester
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Nishio M, Felip E, Orlov S, Park K, Yu CJ, Tsai CM, Cobo M, McKeage M, Su WC, Mok T, Scagliotti GV, Spigel DR, Viraswami-Appanna K, Chen Z, Passos VQ, Shaw AT. Final Overall Survival and Other Efficacy and Safety Results From ASCEND-3: Phase II Study of Ceritinib in ALKi-Naive Patients With ALK-Rearranged NSCLC. J Thorac Oncol. 2020 Apr;15(4):609-617. doi: 10.1016/j.jtho.2019.11.006. Epub 2019 Nov 25. PMID 31778798
- [Derived] Lin YT, Yu CJ, Yang JC, Shih JY. Anaplastic Lymphoma Kinase (ALK) Kinase Domain Mutation Following ALK Inhibitor(s) Failure in Advanced ALK Positive Non-Small-Cell Lung Cancer: Analysis and Literature Review. Clin Lung Cancer. 2016 Sep;17(5):e77-e94. doi: 10.1016/j.cllc.2016.03.005. Epub 2016 Mar 30. PMID 27130468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 105 patients were planned to be enrolled. A total of 124 patients were enrolled and treated with ceritinib.
Period: Overall Study
Arm/Group | LDK378 (Ceritinib)
Started | 124
Discontinued From Treatment Phase | 124
Entered Post-treatment Efficacy f/up | 10
Entered Survival Follow-up | 63
Discontinued From Study | 51
Completed (Completed = discontinued from treatment phase) | 32
Not Completed | 92
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1
Not completed — No longer requires treatment | 1
Not completed — Subject/guardian decision | 2
Not completed — Physician Decision | 6
Not completed — Death | 10
Not completed — Adverse Event | 18
Not completed — Progressive disease | 53

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all patients who received at least one dose of study drug.
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 50
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 74
  Caucasian | 48
  Black | 1
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by Investigator Assessment
Description: ORR per RECIST 1.1 calculated as the percentage of participants with a best overall response (OR) defined as complete response (CR) or partial response (PR) as assessed by the investigator. CR:Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: every 8 weeks (i.e. every 2 cycles; cycle = 28 days), starting from the first day of treatment with LDK378 until permanent discontinuation of study drug up to 5 years
Population: The Full Analysis Set (FAS) consisted of all patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 124
Percentage of participants | 67.7 [58.8 to 75.9]

2. Secondary Outcome: ORR by Blinded Independent Review Committee (BIRC)
Description: ORR per RECIST 1.1 calculated as the percentage of participants with a best overall response (OR) defined as complete response (CR) or partial response (PR) as assessed by BIRC. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: The Full Analysis Set (FAS) consisted of all patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 124
Percentage of participants | 63.7 [54.6 to 72.2]

3. Secondary Outcome: Duration of Response (DOR) as Per Investigator
Description: DOR, calculated as the time from the date of the first documented CR or PR to the first documented progression or death due to any cause, by investigator assessment per RECIST 1.1. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: The set consisted of patients in the Full Analysis Set (FAS) who had confirmed complete response (CR) or partial response (PR) by investigator.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 84
Months | 24.0 [14.8 to 37.5]

4. Secondary Outcome: Duration of Response (DOR) as Per BIRC
Description: DOR, calculated as the time from the date of the first documented CR or PR to the first documented progression or death due to any cause, by BIRC assessment per RECIST 1.1. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: The set consisted of patients in the Full Analysis Set (FAS) who had confirmed complete response (CR) or partial response (PR) as assessed by BIRC.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 79
Months | 27.3 [16.6 to 44.3]

5. Secondary Outcome: Disease Control Rate (DCR) as Per Investigator and BIRC
Description: DCR per RECIST 1.1 is the percentage of participants with best overall response of CR, PR, stable disease (SD) or Non-CR/Non-PD. CR: Disappearance of all non-nodal target lesions. Also, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions that would qualify for PD. PD: At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm.
Time Frame: as for outcome 1
Population: The Full Analysis Set (FAS) consisted of all patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 124
Percentage of participants
  DCR per Investigator | 90.3 [83.7 to 94.9]
  DCR per BIRC | 86.3 [79.0 to 91.8]

6. Secondary Outcome: Time to Response (TTR) as Per Investigator
Description: TTR, calculated as the time from first dose of LDK378 to first documented response (CR+PR), by investigator. This was only on participants with confirmed CR or PR. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: every 8 weeks (i.e. every 2 cycles; cycle = 28 days), starting from the first day of treatment with LDK378 until permanent discontinuation of study drug
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 84
Months | 2.5 (2.66)

7. Secondary Outcome: Time to Response (TTR) as Per BIRC
Description: TTR, calculated as the time from first dose of LDK378 to first documented response (CR+PR), by BIRC assessment. This was only on participants with confirmed CR or PR. CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 79
Months | 2.2 (1.22)

8. Secondary Outcome: Overall Intracranial Response Rate (OIRR) as Per Investigator
Description: OIRR calculated as the ORR (CR+PR) of lesions in the brain for patients who have measureable disease in the brain at baseline by investigator.
Time Frame: as for outcome 1
Population: The set consisted of patients in the Full Analysis Set (FAS) who had measurable target lesions in brain at baseline by investigator.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 10
Percentage of participants | 20.0 [2.5 to 55.6]

9. Secondary Outcome: Overall Intracranial Response Rate (OIRR) as Per BIRC
Description: OIRR calculated as the ORR (CR+PR) of lesions in the brain for patients who have measureable disease in the brain at baseline by BIRC.
Time Frame: as for outcome 1
Population: The set consisted of patients in the Full Analysis Set (FAS) who had measurable target lesions in brain at baseline by BIRC.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 13
Percentage of participants | 61.5 [31.6 to 86.1]

10. Secondary Outcome: Progression-free Survival (PFS) Per Investigator and BIRC
Description: PFS, defined as time from first dose of LDK378 to progression or death due to any cause, as assessed by investigator and BIRC assessments.
Time Frame: as for outcome 1
Population: The Full Analysis Set (FAS) consisted of all patients who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 124
Months
  PFS per Investigator | 16.6 [11.0 to 23.2]
  PFS per BIRC | 19.4 [10.9 to 29.3]

11. Secondary Outcome: Overall Survival (OS)
Description: OS, defined as time from first dose of LDK378 to death due to any cause
Time Frame: Time from the date of first dose of LDK378 to the date of death due to any cause up to 5 years
Population: The Full Analysis Set (FAS) consisted of all patients who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | LDK378 (Ceritinib)
Number analyzed (Participants) | 124
Months | 51.3 [42.7 to 55.3]

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 5 years.
Groups:
- LDK378 Ceritinib): Participants on this arm took oral LDK378 750 mg once daily.
Arm/Group | LDK378 Ceritinib)
All-Cause Mortality (participants affected / at risk) | 56/124
Serious Adverse Events (participants affected / at risk) | 50/124
Other Adverse Events (participants affected / at risk) | 123/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDK378 Ceritinib) (N=124)
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 4
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anal inflammation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Oesophageal stenosis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 1
Fatigue (General disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 2
Hepatitis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 4
Nosocomial infection (Infections and infestations) | 1
Parvovirus infection (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Post procedural infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Weight decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diabetic ketosis (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chordoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 2
Cognitive disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Radicular pain (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDK378 Ceritinib) (N=124)
Anaemia (Blood and lymphatic system disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 11
Abdominal distension (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 51
Abdominal pain upper (Gastrointestinal disorders) | 19
Constipation (Gastrointestinal disorders) | 35
Diarrhoea (Gastrointestinal disorders) | 106
Dyspepsia (Gastrointestinal disorders) | 15
Gastrointestinal pain (Gastrointestinal disorders) | 9
Haemorrhoids (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 97
Stomatitis (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 89
Asthenia (General disorders) | 19
Chest discomfort (General disorders) | 9
Fatigue (General disorders) | 47
Malaise (General disorders) | 9
Non-cardiac chest pain (General disorders) | 19
Pyrexia (General disorders) | 23
Influenza (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 18
Pneumonia (Infections and infestations) | 8
Upper respiratory tract infection (Infections and infestations) | 25
Urinary tract infection (Infections and infestations) | 10
Alanine aminotransferase increased (Investigations) | 65
Amylase increased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 58
Blood alkaline phosphatase increased (Investigations) | 29
Blood creatinine increased (Investigations) | 33
Creatinine renal clearance decreased (Investigations) | 8
Electrocardiogram QT prolonged (Investigations) | 20
Gamma-glutamyltransferase increased (Investigations) | 36
Lipase increased (Investigations) | 9
Weight decreased (Investigations) | 47
Weight increased (Investigations) | 8
White blood cell count decreased (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 69
Hyperglycaemia (Metabolism and nutrition disorders) | 15
Hyperkalaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 14
Hyponatraemia (Metabolism and nutrition disorders) | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 25
Back pain (Musculoskeletal and connective tissue disorders) | 32
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 21
Headache (Nervous system disorders) | 31
Paraesthesia (Nervous system disorders) | 8
Insomnia (Psychiatric disorders) | 11
Dysuria (Renal and urinary disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 15
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 18
Rash (Skin and subcutaneous tissue disorders) | 28
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2015-12-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT01685138/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT01685138/SAP_001.pdf